CLINICAL TRIAL: NCT02713503
Title: HFCV Mobile Device Vehicle Integration Assessment
Brief Title: Evaluating Electronic Devices in a Driving Simulator
Status: Completed | Type: Observational
Sponsor: Clemson University (Other)
Collaborators: National Highway Traffic Safety Administration (NHTSA) (U.S. Federal Agency); Westat (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-167
Record Dates: First submitted 2016-02-12; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Drivers: Driving Observation and VisionCoach
  Interventions: Other: Driving Observation; Other: VisionCoach

INTERVENTIONS:
Other: Driving Observation — Driving observation using the DriveSafety CDS-250 Driving Simulator.
Other: VisionCoach — Visual field evaluation using VisionCoach

SUMMARY:
The purpose of this study is to evaluate a variety of technologies in a driving simulator. Specifically, this research will provide a direct comparison of driver performance measures under various modes of mobile device interaction.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate a variety of technologies in a driving simulator. Specifically, this research will provide a direct comparison of driver performance measures under various modes of mobile device interaction. The study will be conducted at CU-ICAR using the DriveSafety CDS-250 driving simulator. The experiment will be a key step in understanding what driver performance challenges and errors may occur under various interaction modes in the driving context. Results will investigate differences in driving performance in the presence and absence of full device pairing with vehicle electronics and what criteria might be considered for proposed pairing requirements. The driving simulator tasks will focus on visual scanning ability while engaging in secondary tasks using mobile devices such as (but not limited to) handheld phones with and without Bluetooth, mounted touchscreen displays, various voice-based interfaces, and the novel display system. Tasks will include activities such as making voice calls, text messaging, searching for points of interest on maps, and traditional in-vehicle activities such as changing the temperature, fan speed, radio station, etc. The number of tasks and interaction modes will vary between participants with up to 6 modes included per participant (e.g. handheld, mounted ipad, voice control).

The technologies will be integrated with the DriveSafety CDS-250 driving simulator. Participants will complete the Functional Object Detection (FOD) visual scanning task that requires a driver to maintain lane position, respond to brake events in the central field of view, and respond to target events that appear in the periphery. In addition, participants will be asked to concurrently complete the mobile-device tasks using the interaction modes described previously and occasionally respond to notifications simulating connected-vehicle interactions. Primary outcomes will include driving performance (lane tracking and speed maintenance), FOD peripheral task performance (% identified, response time), FOD braking task performance (% identified, response time, false positive responses), and subjective measures including workload, interface preferences, and open ended items describing their reactions to each interface.

Participants will complete training to get comfortable driving the simulator while driving on a straight road and then repeat the task using the cruise control prior to driving the experimental conditions. Participants will be recruited by word of mouth as well as through the use of flyers, newspaper advertisements, and talks in the community. All data will be collected in the driving simulator lab at CU-ICAR. We plan to share the findings of this research with designers, practitioners and researchers at conferences and through academic publications.

Participants will complete a vision screening using a standard eye chart and will complete a visual scanning task using an interactive light board where the participants will stand (or sit) in front of a board with moving lights and asked to identify the locations, colors, letters and numbers of the lights by pressing their location on the board.

DriveSafety™ CDS-250 Driving Simulator The CDS-250 driving simulator is designed as a rehabilitation tool which occupies a smaller footprint than traditional driving simulators. The simulator has a partial cab consisting of an adjustable driver's seat, center console, instrument cluster, and standard vehicle controls (steering wheel, accelerator, brake). Two input buttons are located on the steering wheel in the "3:00" and "9:00" positions. The display consists of three 19" (diagonal) LCD screens each with a resolution of 1440 X 900 pixels. The left and right screens are each rotated 30 degrees off-plane from the center screen toward the driver. The total horizontal width of this display configuration is 49". In addition to using the driving simulator for driving related tasks, a variety of reaction time tasks have been developed to work on patients' coordinated muscle movements, information processing, and reaction times.

ELIGIBILITY:
Inclusion Criteria:

* Licensed drivers who are over the age of 18 who meet the SC vision screening of 20/40

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy drivers
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2013-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Driving performance as assessed by lane tracking (5 discrete categories that correspond with lane positioning) | 1 day
Driving performance as assessed by speed maintenance (mean, range and variation of driver speed) | 1 day

SECONDARY OUTCOMES:
Functional Object Detection peripheral task performance as assessed by detect and respond to stimuli in the drivers periphery | 1 day
Functional Object Detection braking task performance as assessed by detect and respond to stimuli by button pressing or braking | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Johnell Brooks, PhD, Principal Investigator — Clemson University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brooks J, Seeanner J, Hennessy S, Manganelli J, Crisler M, Rosopa P, Jenkins C, Anderson M, Drouin N, Belle L, Truesdail C, Tanner S. Interactive Tools for Measuring Visual Scanning Performance and Reaction Time. Am J Occup Ther. 2017 Mar/Apr;71(2):7102350010p1-20102350020p6. doi: 10.5014/ajot.2017.020461. PMID 28218598